CLINICAL TRIAL: NCT00671801
Title: Phase I Trial of Irinotecan Plus Lenalidomide in Adult Patients With Recurrent Glioblastoma Multiforme
Brief Title: Irinotecan Plus Lenalidomide in Adult Patients With Recurrent Glioblastoma Multiforme: Phase I
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Toxicity
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0472; NCI-2012-01684 (Registry Identifier: NCI CTRP); NCT02369367 (obsolete NCT alias)
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Malignant Gliomas
Keywords: Malignant Gliomas; Glioblastoma Multiforme; Gliosarcoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma; Camptosar; Irinotecan; CPT-11; Lenalidomide; Revlimid; CC-5013
MeSH Terms: conditions — Glioma; Glioblastoma; Gliosarcoma; Astrocytoma; Oligodendroglioma | interventions — Irinotecan; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Irinotecan + Lenalidomide (Experimental): Irinotecan 200 mg/m^2 intravenous once every 2 weeks on days 1 and 15; Lenalidomide orally 7.5 mg/day on Cycle 1 Days 1-21 and 10 mg/day on Cycle 2 Days 1-21.
  Interventions: Drug: Irinotecan; Drug: Lenalidomide

INTERVENTIONS:
Drug: Irinotecan — 200 mg/m^2 by vein over 90 minutes once every 2 weeks on days 1 and 15.
  Other Names: Camptosar; CPT-11
Drug: Lenalidomide — Given orally at escalating doses beginning 7.5 mg/day on Cycle 1 Days 1-21 and 10 mg/day on Cycle 2 Days 1-21.
  Other Names: Revlimid; CC-5013

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of lenalidomide combined with Camptosar (irinotecan) as well as to see if this drug combination can help control malignant gliomas.

Researchers will also study if a special magnetic resonance imaging (MRI) technique (dynamic MRI scan) is useful in looking at the effect of treatment on the tumor. Another goal is to learn the effect of lenalidomide on tumor tissue in patients who need surgery for the disease.

DETAILED DESCRIPTION:
Lenalidomide is designed to change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. Therefore, in theory, it may decrease or prevent the growth of cancer cells.

Irinotecan is designed to stop cancer cells from dividing by causing "breaks" in the tumor cell DNA (the genetic material of cells), which may cause the cancer cells to die.

There are 2 parts to this study. In the first part (Phase I) of this study, researchers will try to find the highest tolerable dose of the study drug combination. In the second part (Phase II) of this study (after the highest tolerable dose is reached), researchers will try to learn the effectiveness of the study drug combination. If you are found to be eligible to take part in this study, you will be enrolled in Phase I or Phase II depending on which part is open at the time.

Phase I:

For this phase, you will be enrolled in a group of at least 3 participants to begin receiving lenalidomide and irinotecan. The dose of the study drug combination you receive will depend on when you enrolled in this study. At each dose level, if no intolerable side effects occur (after 4 weeks), the next 3 participants will be enrolled to receive a higher dose of the study drug combination. This process will continue until the highest tolerable dose of the study drug combination is reached. You will remain on the same dose throughout this study.

You will take lenalidomide by mouth (capsules) every morning on Days 1-21 of each 28 day cycle. Swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules. In addition, you will also receive 1 additional dose of lenalidomide by mouth before the beginning of Cycle 1 (on Day 0 of Cycle 1).

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose). If you take too much lenalidomide or overdose, call your study doctor or health care provider or poison control center right away.

You will receive irinotecan by vein over 90 minutes once every 2 weeks (on Days 1 and 15). One cycle of treatment is 28 days long. You will have a "rest" period on Days 22-28 where you will not receive any study treatment.

Phase II:

For this phase, you will take lenalidomide by mouth (capsules) every morning on Days 1-21. Swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose). If you take too much lenalidomide or overdose, call your study doctor or health care provider or poison control center right away.

You will receive irinotecan by vein over 90 minutes once every 2 weeks on Days 1 and 15. One cycle of treatment is 28 days long. You will have a "rest" period on Days 22-28 where you will not receive any study treatment.

Some participants in the Phase II study may also qualify for a component (a subset) of this study that will enroll up to 10 participants who will be undergoing surgical resection (removal of all or part of tissue) of the tumor. If the MRI scan (done during screening) shows that you have tumor regrowth and your doctor has recommended surgery to remove the regrown tumor, you will be eligible for this subset of the study.

For the subset, you will take lenalidomide (in the same manner as mentioned above), before surgery, for 3 days in a row with the last dose to be taken on the day of surgery.

Blood (about 2 teaspoons) will be drawn for pharmacokinetic (PK) testing on the first and second days that you take the study drug before surgery and on the day of surgery. PK testing measures the amount of study drug in the body at different time points.

Also, leftover tumor tissue (removed during your surgery) will be collected and used for testing to learn the effect of lenalidomide on your tumor tissue. The leftover tumor tissue samples will also be stored for research tissue/blood bank after the last participant completes the study. You will have a standard MRI scan and a dynamic MRI scan within 3 days after surgery.

Before your leftover tumor tissue samples can be used for research, the people doing the research must get specific approval from the Institutional Review Board (IRB) of M. D. Anderson. The IRB is a committee made up of doctors, researchers, and members of the community. The IRB is responsible for protecting the participants involved in research studies and making sure all research is done in a safe and ethical manner. All research done at M. D. Anderson, including research involving your leftover tumor tissue samples from this bank, must first be approved by the IRB.

All participants:

During treatment, you will have a complete physical exam and brain and spinal exam (performed by checking your coordination and strength by looking at how you walk and pull objects), which will be done every one cycle if you are in Phase I and every 2 cycles if you are in Phase II. On Day 1 of every cycle you will discuss birth control methods. You will have blood drawn (about 2 teaspoons each time) for routine tests once a week during Cycle 1 and then every 2 weeks in further cycles. You will have blood drawn (about 2 teaspoons each time) for routine tests on Day 15 of Cycle 1 and then on Day 1 in further cycles (every one cycle if you are in Phase I and every 2 cycles if you are in Phase II). You will also have a dynamic MRI scan done every 2 cycles after completion of Cycle 2. For all women who are able to have children: You will have a pregnancy test performed by your doctor within 10 - 14 days and 24 hours prior to starting lenalidomide therapy, even if you have not had any menses due to treatment of your disease or had as little as one menstrual period in the past 24 months. If you have regular or no menstrual cycles, you will have pregnancy tests every week for the first 28 days, then every 28 days while taking lenalidomide, when you stop taking lenalidomide, then 28 days after you have stopped taking lenalidomide. If you have irregular menstrual cycles, you will have pregnancy tests every week for the first 28 days, then every 14 days while taking lenalidomide, again when you have been taken off of lenalidomide therapy, and then 14 days and 28 days after you have stopped taking lenalidomide.

Treatment on this study will continue for at least 1 year, as long as the tumor does not grow back and there are no intolerable side effects. Treatment beyond 1 year will be based on whether the study doctor thinks that you may benefit without severe side effects.

If at any time during treatment the disease gets worse or you experience any intolerable side effects, you will be taken off this study, and your study doctor will discuss other treatment options with you.

Once you are completely off this study for any reason, you will have an end-of-study visit. During this visit, you will have a complete physical exam, including measurement of your height and weight. You will be asked how well you are able to perform the normal activities of daily living (performance status evaluation). You will have a brain and spinal exam. You will have blood drawn (about 5 teaspoons) for routine tests. This routine blood draw will include a pregnancy test for women who are able to have children. About 1 teaspoon of blood will be drawn to test for the ability of your blood to clot normally.

PK and Biomarker testing for Phase I:

If you are in Phase I, the following tests and procedures will be performed:

* Blood (about 1 teaspoon each time) will be drawn 6 times per day on Days 0, 1, and 4 of Cycle 1 for PK testing.
* Blood (about 1 teaspoon each time) will be drawn 3 times per day on Days 0, 1 and 4 of Cycle 1, and 1 time on Day 1 of Cycle 2 for biomarker testing. Biomarkers are chemical "markers" in the blood and/or tissue that may be related to your reaction to the study drug.
* If you experience a skin rash due to an intolerable dose of the study drug, a punch biopsy of your skin will be performed on a rash area of your body. This tissue will be used for testing to help the doctors understand what caused the serious reaction and for biomarker testing. To perform a punch biopsy, a hollow knife tool is used to remove a small coin-shaped sample of tissue.

This is an investigational study. Lenalidomide and irinotecan are FDA approved and commercially available for the treatment of some cancers. Their combination use is investigational and authorized for use in research only. Up to 51 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven World Health Organization (WHO) grade III and IV malignant gliomas will be eligible for the phase I portion of this study. For the Phase II part, patients with histologically proven supratentorial WHO grade IV malignant glioma (Glioblastomas (GBM) and gliosarcoma) will be eligible
2. There must be unequivocal evidence for tumor recurrence or progression by MRI scan and the patient must have received radiation therapy previously.
3. Patients must be capable of understanding and voluntarily signing an informed consent form.
4. Age >/=18 years at the time of signing the informed consent form.
5. Karnofsky performance status of >/=60 at study entry
6. Able to adhere to the study visit schedule and other protocol requirements.
7. For the phase I portion of the study, patients may have any number of prior relapses provided all other eligibility criteria, particularly the functional status, are met.
8. (7. continued) For the phase II portion of the study, no more than 2 prior relapses are allowed. Patients must have failed prior radiation therapy and in order to exclude the possibility of radiological pseudoprogression for patients with GBM, must have an interval >/= 12 weeks from the completion of chemoradiation therapy to the study entry unless tumor progression has been confirmed by either surgery or by appropriate imaging studies (eg. PET scan, MR Spectroscopy etc). Tumor regrowth after chemoradiation followed by adjuvant chemotherapy is considered one relapse.
9. The baseline on-study MRI should be performed within 14 days prior to registration and on a steroid dosage that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and the initiation of therapy (or at that time), a new baseline MRI is required. The same type of scan, i.e., MRI, must be used throughout the period of protocol treatment for tumor measurement.
10. Patients must have recovered from the toxic effects of prior therapy: 4 weeks from any investigational agents, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, cis-retinoic acid, etc. (radiosensitizer does not count).
11. ( 10. continued) Patients who receive irinotecan for non-therapeutic purposes unrelated to this study (such as presurgically for obtaining pharmacology data for the agent) will be eligible to enter the study provided they have recovered from the toxic effects of the agent if any. Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
12. Laboratory test results within these ranges: 1) Absolute neutrophil count >/= 1.5 x 10^9/L. 2) Platelet count >/= 100 x 10^9/L. 3) Serum creatinine </= 1.5 mg/dL. 4) Total bilirubin </= 1.5 mg/dL. 5) aspartate aminotransferase (AST/SGOT) and alanine transaminase (ALT/SGPT) </= 2 x upper limit of normal (ULN).
13. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.
14. (13. continued) FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
15. Disease free of prior malignancies for >/= 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in-situ" of the cervix or breast.
16. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender.
17. There must be unequivocal evidence for tumor recurrence or progression by MRI scan (Phase II surgical, pre-operative)
18. Ability to obtain sufficient tumor specimen for the performance of the biomarker studies in the opinion of the treating physician and surgeon (Phase II surgical, pre-operative)
19. Meets all the inclusion/exclusion criteria for the phase II study except patients are not required to be on a stable dose of steroids prior to surgery.(Phase II surgical, pre-operative)
20. Patient must meet the pre-entry pregnancy testing and birth control requirement prior to the first pre-operative dose of lenalidomide (Phase II surgical, pre-operative)
21. The patient has consented to the surgical resection and correlative lab evaluations (phase II surgical, pre-operative)
22. Post-operative MRI scan performed no later than 96 hours and on a stable or reducing dose of steroids. (if treatment begins more than 14 days after the 96 hour scan, a new MRI scan including dynamic contrast-enhanced (DCE) MRI if there is residual tumor will be required to serve as the baseline MRI for efficacy analysis) (Phase II surgical, post-operative)
23. Must have recovered from the effects of surgery. (phase II surgical, post-operative)
24. Must have confirmation of recurrent tumor by pathology criteria.(phase II surgical, post-operative)
25. The patient has followed the on study requirements for birth control and pregnancy testing since the initial pre-operative dose of lenalidomide. (phase II surgical, post-operative)
26. The post operative complete blood count (CBC) and chemistry panel meet the entry criteria # 12.
27. The patient continues to meet all the inclusion/exclusion criteria of the study outlined above except inclusion criteria #9. (phase II surgical, post-operative)
28. Able to take warfarin or use low molecular weight heparin for the duration of study treatment
29. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent.
2. Pregnant or breast feeding females.
3. Any condition, including the presence of clinically significant laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study. These would include a) Active infection(including persistent fever) b) Diseases or conditions that obscure toxicity or dangerously alter drug metabolism c) Serious intercurrent medical illness (e.g.symptomatic congestive heart failure).
4. Known hypersensitivity to thalidomide or lenalidomide.
5. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
6. Prior recurrence with irinotecan - (prior treatment with lenalidomide as single agent is permitted). Patients who have received irinotecan for non-therapeutic purposes (for eg., as part of a pharmacology study without therapeutic intent) will remain eligible for enrollment into the study. Patients who have received thalidomide or lenalidomide not in combination with irinotecan or other cytotoxic agents remain eligible for enrollment into the study.
7. Concurrent use of other anti-cancer agents or treatments.
8. No exclusion to this study will be based on race. Minorities will actively be recruited to participate. The malignant glioma patient population treated at MD Anderson Cancer Center over the past year is as follows: 1) American Indian or Alaskan Native - 0. 2) Asian or Pacific Islander - <2%. 3) Black, not of Hispanic Origin - 3%. 4) Hispanic - 6%. 5) White, not of Hispanic Origin - 88%. 6) Other or Unknown - 2%. Total-100%
9. Patients must not be on enzyme inducing anticonvulsants; if the treating physician elects to change the medication to a non-enzyme inducing agent, a 1-week wash out period will be required after stopping Enzyme-Inducing Anti-Epileptic Drugs (EIAED) prior to initiation of irinotecan.
10. In the phase II portion of the study, prior antitumor treatment with bevacizumab is not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04-29 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Lenalidomide and Irinotecan | First cycle (28 days)
  MTD declared dose level if </= 1 dose limiting toxicity (DLT) occurs.

CONTACTS AND LOCATIONS:
Overall Officials: John DeGroot, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org